CLINICAL TRIAL: NCT04743544
Title: Influence of CYP2C19 Genotype on Safety and Efficacy of Voriconazole in Pediatric Patients With Hematologic Malignancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Principal Investigator, Mukaddes Gumustekin, Full Professor, Dokuz Eylul University
Other Study IDs: 19-AKD-124
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Adverse Drug Reactions
Keywords: voriconazole; invasive aspergillosis; CYP2C19 polymorphisms; pharmacogenetics; hematologic malignancy; pediatric population; efficacy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Hematologic Neoplasms | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 mL of blood sample collected into an EDTA (Ethylenediaminetetraacetic Acid) tube for PGx analysis and another 2 mL of blood sample collected into an EDTA (Ethylenediaminetetraacetic Acid) tube for voriconazole TDM
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Voriconazole: All eligible patients will be followed up for voriconazole related adverse drug events and efficacy
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — This is an observational study and only the patients already on voriconazole treatment will be included in the study.

SUMMARY:
Voriconazole is a drug used to treat invasive fungal infections. The amount of voriconazole in a person's blood helps to determine how effectively it treats an infection, and how safe it is. Patients respond differently when receiving the same dose - some clearly benefit, other patients experience side effects, and others see limited improvement in their infection.

Voriconazole is broken down in the liver mainly by an enzyme called CYP2C19, before being excreted from the body. The activity of CY2C19 differs between people because of variation in the DNA that encodes the body's instructions to make CYP2C19.

If CYP2C19 activity is very high, voriconazole blood levels may remain below the target range when a patient receives a standard dose of voriconazole, which may be insufficient to treat their infection. Besides, children tend to have faster voriconazole metabolism regardless of the genetic makeup, mainly because of higher liver mass/body proportion. That's why, younger patients needs higher doses and it is harder for them to reach target range. Having a high CYP2C19 activity and being young combined may cause to consider choosing an alternative drug. By contrast, decreased CYP2C19 activity due to genetic variation may result in excessively high voriconazole blood levels, predisposing to serious side effects.

Therefore, knowing a patient's CYP2C19 genetic makeup is very important for predicting their response to voriconazole.

Thus, we aim to determine the influence of genetic variation in CYP2C19 on the frequency and severity of side effects related to voriconazole, and on the effectiveness of voriconazole for treating serious fungal infections. The findings from this study will contribute to determining the optimal dose of voriconazole that patients with different genetic variants in CYP2C19 should be started on, and will take us one step closer to both understanding the genetic structure of CYP2C19 in the Turkish population, and to 'personalised medicine'.

DETAILED DESCRIPTION:
Invasive fungal infections are the leading cause of mortality and morbidity in immune compromised children. Aspergillus species are reported to be the most common molds that cause invasive infections among pediatric patients both in the United States and in Europe.

Voriconazole is recommended as the first line therapy for invasive Aspergillosis. The major proportion of the drug undergoes hepatic metabolism via cytochrome enzymes. The hepatic cytochrome enzyme that mainly involves in the metabolism of voriconazole is CYP2C19, which is known to be highly polymorphic. So far, more than 30 variant alleles have been defined in the gene that codes CYP2C19 enzyme.

Polymorphisms in CYP2C19 gene are associated with alterations in voriconazole metabolism. It is postulated that only 35-50% of the populations has normal metabolic activity for this drug. The carriers of defective alleles (*2/*2, *2/*3, *3/*3) in CYP2C19 gene have slower metabolic activity for voriconazole, while the carriers of *17 allele have increased enzyme activity and higher metabolic capacity for the drug.

Voriconazole has a narrow therapeutic window. When the therapy is initiated with standard doses, interpersonal differences in CYP2C19 activity make it difficult to remain in the optimal therapeutic range. Furthermore, it is reported that voriconazole concentrations in pediatric patients can exhibit up to 3-fold variation among individuals and it is extremely hard to reach and remain therapeutic concentration in younger children. As low serum concentrations cause decreased efficacy, supratherapeutic concentrations may cause voriconazole toxicity which also leads to significant morbidity, mortality and high treatment costs.

To ensure desired efficacy and safety of voriconazole treatment, therapeutic drug monitoring (TDM) is recommended, but unfortunately, it is not a part of routine clinical care in many hospitals, due to frequent blood sampling and analysis requirements and the high analysis costs. On the other hand, starting the therapy with standard doses and adjusting it with subsequent TDMs may cause delay in selecting optimal voriconazole dose and providing effective treatment.

It is reported that, pediatric patients those are initiated voriconazole therapy with pharmacogenetic-guided dose selection reaches targeted serum voriconazole concentration 4-fold faster than the patients those are given standard doses and undergoes subsequent dose adjustments according to TDM results. Thus, CYP2C19 genotyping is essential in reaching the optimal voriconazole concentration in shorter times. Genotype-guided first dose selection would make it easier to reach the targeted serum voriconazole concentration, minimize frequent TDM requirement, prevent the treatment failure and lead to better clinical outcomes. On the other hand, pharmacogenetic analysis results can also be used for adjusting dose of other drugs that is metabolized by the same enzyme.

We could only located one conference proceeding reporting the effect of CYP2C19 polymorphisms on safety of voriconazole use in 6 patients in Turkish population. Current literature is limited and the guidelines does not make a clear recommendation about the pharmacogenetic-guided dose selections. Thus, to build safe pharmacogenetic- guided dose selection algorithms, more data in that field is required.

This study is designed to prospectively determine the influence of CYP2C19 polymorphisms on frequency and severity of voriconazole related adverse event reactions during the study follow up period and on the efficacy of voriconazole treatment/ prophylaxis. Samples for pharmacogenetic analysis will be stored for further studies depending on participant's and the parents' discreation.

METHOD This is a multi centre, observational cohort study.

Study population:

Patients aged between ≥2 years and <18 years hospitalized in pediatric hematology clinics in research centers (Dokuz Eylul University Hospital, Ege University Hospital, Izmir University of Health Sciences Tepecik Training and Research Hospital) due to a hematological malignancy (acute lymphoblastic leukemia, acute myeloid leukemia) and receiving voriconazole as part of invasive fungal infection prophylaxis or treatment.

Data and sample collection 1.1.1.Data collection: At baseline, demographics and clinical information will be recorded from all patients directly and complemented from their medical records. All patients will be followed up by the research team daily for the first 7 days following voriconazole initiation, and then on days 14, 30 and 60. All follow up will be initially via assessment of medical records, with additional data input from the patient directly. The medical records include: the electronic hospital record system (PROBEL), paper-based patient records and other patient follow-up- documents.

During routine clinical care, ADRs are monitored daily by a pediatric hematology fellow and/or pediatrician. On days one to seven following voriconazole initiation, the investigators will record these clinical evaluations daily; they will also capture these data on days 14 and 30.

For participants that had either started voriconazole active treatment before they were recruited, or were recruited during the maintenance phase of their voriconazole regimen, the research team will assess their medicals records retrospectively between the point of recruitment and day one of their active voriconazole treatment to detect ADRs.

On days 30 and 60, patient survival will be recorded by review of patient records only.

Treatment response (efficacy) will be determined based on the EORTC/MSG consensus criteria. These data will be obtained at all follow up points (from day one to seven, and days 14, 30 and 60).

1.1.2.Sample collection: 1.1.2.1.Samples fo PGx analysis: All pediatric patients with a hematologic malignancy (acute lymphoblastic leukemia, acute myeloid leukemia) hospitalized aforementioned study centers and their parents will be informed of the study. Those agree to participate in will donate 2 mL blood sample collected into an EDTA (Ethylenediaminetetraacetic Acid) tube on day one whilst blood samples are being taken from the patient for daily routine clinical purposes (without requiring any other needle insertion). Samples for PGx analysis will be coded and stored securely in Dokuz Eylul University Hospital, Department of Medical Pharmacology. The samples will be stored -80 celcius degree until used up. PGx analysis will be performed in the Department of Medical Genetics at Dokuz Eylul University Hospital at the end of the study. Participants and physicians will not be informed of the participant's genotype during the study period. The participant's clinical care will not be affected in any way by taking part in the study.

1.1.2.2.Samples for voriconazole concentration determination: The patients those start using voriconazole as part of invasive fungal infection prophylaxis or treatment will The second 2 mL blood sample will be collected into a red cap tube on the fifth day (9th dose) of treatment before the morning voriconazole dose, again whilst blood is being collected as part of routine clinical care (without requiring any other needle insertion) to determine the trough voriconazole concentration at steady state. This blood sample will be centrifuged and the serum stored in the Department of Medical Pharmacology at the Dokuz Eylul University Faculty of Medicine. When follow up is completed for a given patient, this serum sample will be transferred to an accredited laboratory in Istanbul, Turkey, with maintenance and assurance of the cold chain during sample transportation to guarantee sample integrity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between ≥2 years and <18 years
* Receiving voriconazole for the treatment of an invasive fungal infection (IFI) and are within the first five days of the treatment course, OR are receiving voriconazole for the secondary prophylaxis against IFI during or after chemotherapy
* Agree to give one additional blood sample twice during the study for the purposes of pharmacogenetic analysis and determination of the serum trough voriconazole concentration, whilst their blood is being collected during normal clinical follow up without the requirement for any additional intravenous intervention
* Are willing and able to give informed consent and sign the informed consent form (by the patients and the parents OR the legal guardians)

Exclusion Criteria:

* Have previously had CYP2C19 PGx testing performed
* Pregnant/breastfeeding
* Have cognitive impairment and/or psychiatric disorders and/or any other condition that will draw into question their capacity to provide informed consent
* Have severe hepatic insufficiency (Child-Pugh Class C) and have renal failure (estimated GFR <15ml/min /1,73m2)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged between ≥2 years and <18 years hospitalized in pediatric hematology clinics in research centers (Dokuz Eylul University Hospital, Ege University Hospital, Izmir University of Health Sciences Tepecik Training and Research Hospital) due to a hematological malignancy (acute lymphoblastic leukemia, acute myeloid leukemia) and receiving voriconazole as part of invasive fungal infection prophylaxis or treatment.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of voriconazole related adverse drug reactions | Follow up period for primary outcome is 30 days for each participant
  Voriconazole related adverse drug reactions of grade 3-5 systematically evaluated using Liverpool Causality Assessment Tool identified during study follow up.
  Severity of all adverse events will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

SECONDARY OUTCOMES:
Non-response to voriconazole | Follow up period for this outcome is 60 days for each participant
  The efficacy of voriconazole treatment will be assessed based on reviews of clinical, mycological and radiological data according to the Mycoses Study Group and European Organization for Research and Treatment of Cancer Consensus Criteria (EORTC/MSG criteria).
Voriconazole trough concentration | 30 minutes before the 9th dose of voriconazole
  Voriconazole trough concentration will be measured once for each participant from plasma samples collected 30 minutes before the 9th dose of voriconazole
Survival | On days 30 and 60
  Patient survival will be evaluated on days 30 and 60 by reference to the Dokuz Eylul University Hospital Hematology Service; date of death will be captured to permit survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mukaddes Gumustekin, Professor, MD, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided